CLINICAL TRIAL: NCT07094841
Title: Comparative Study Between The Effect of Three Dimensional Printed Appliances Herbst and Mandibular Anterior Repositioning Appliance (MARA) on Posterior Airway Space And Temporomandibular Joint TMJ in Growing Class II Malocclusion Patients (Randomized Clinical Trial)
Brief Title: Comparative Study Between Two 3D Functional Appliances Herbst and Mandibular Anterior Repositioning Appliance (MARA) on Posterior Airway Space And TMJ in Growing Class II Malocclusion Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moataz Sleem Ahmed Ali (Other)
Responsible Party: Sponsor-Investigator, Moataz Sleem Ahmed Ali, Master's degree candidate in orthodontics, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3D Herbst Mara- c2 RCT 2025
Record Dates: First submitted 2025-07-15; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mal Occlusion Class 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- herbst group (Experimental)
  Interventions: Device: 3D PRINTED herbst appliance
- mara group (Experimental)
  Interventions: Device: 3d printed mara

INTERVENTIONS:
Device: 3D PRINTED herbst appliance — participants will receive treatment with herbst appliance for 4 to 5 months
  Arms: herbst group
Device: 3d printed mara — participants will receive treatment with mara appliance for 4 to 5 months
  Arms: mara group

SUMMARY:
The aim of this study is to evaluate effect of three dimensional printed appliances Herbst appliance and Mandibular Anterior Repositioning Appliance (MARA) on Posterior Airway Space (PAS) and Temporomandibular Joint (TMJ) in growing patients with Class II malocclusion.

Primary outcome:

Effect of three dimensional printed appliances Herbst appliance and Mandibular Anterior Repositioning Appliance (MARA) on Class II malocclusion in growing patients.

Secondary outcome: To evaluate effects of two different three dimensional printed functional appliances on Posterior Airway Space (PAS) and Temporomandibular Joint (TMJ).

DETAILED DESCRIPTION:
Class II malocclusion is the most common sagittal skeletal imbalance. It can result from mandibular retrusion, maxillary overgrowth, or a posteriorly positioned glenoid fossa According to McNamara (1981), mandibular skeletal retrusion is the predominant skeletal feature in Class II cases, while maxillary skeletal protrusion is relatively uncommon. Class II malocclusion frequently includes Mandibular retrusion, protruding maxillary incisors, increased overjet, imperfect lip closure, and a higher risk of dental trauma and functional disruptions.

Functional appliances aim to correct functional habits, prevent trauma to protrusive incisors, improve facial esthetics, and stimulate mandibular growth for better occlusal balance and long-term stability during development.

Their primary objective is to stimulate mandibular growth by advancing the mandible into a Class I occlusal relationship, and the expectation is that the condylar processes will remodel superiorly and posteriorly in the condylar fossae. Functional appliances are used during growth.They are classified as removable or fixed, with fixed types including rigid, hybrid, and flexible designs. Studies have indicated that rigid fixed functional appliances yield the most effective results in growing patients.

Patient compliance is a critical factor influencing the effectiveness of functional appliances. so, it is important to evaluate removable and fixed appliances separately to accurately assess their clinical efficacy and identify any differences in treatment outcomes. The mandibular anterior repositioning appliance (MARA) is a functional device used to correct Class II malocclusion by repositioning the mandibular condyles anteriorly and inferiorly, promoting remodeling of the condyles and temporal fossae.

The Herbst appliance is a rigid fixed functional device used for Class II correction and is effective over a short treatment period of six to eight months. It functions as an artificial joint by advancing the mandible forward, inducing a "bite-jumping" effect. it has been shown to produce stable and favorable dentoskeletal effects in the correction of Class II malocclusion Additive manufacturing (AM) is a technique for producing three-dimensional (3D) objects by layering materials. Initially introduced in 1980, the process begins with a 3D design that is sliced into cross sections and transmitted to a 3D printer.. This technology is widely applied in medical fields, such as dental and orthodontic appliances. The posterior airway space (PAS), located between the posterior pharyngeal wall and the base of the tongue or soft palate, is part of the extrathoracic airway. A reduced PAS is linked to conditions such as obstructive sleep apnea (OSA) and snoring, Mandibular hypoplasia can present with a range of clinical symptoms, from minor aesthetic concerns to functional impairments and OSA.

The temporomandibular joint (TMJ) is a complex joint that facilitates mandibular movement and adapts structurally in response to external factors such as age, muscle activity, and occlusal forces.

This study aims to explore and compare the impact of these two 3D-printed appliances on the posterior airway space and TMJ structures, providing insight into their relative effectiveness in improving both skeletal and functional outcomes during growth modification

ELIGIBILITY:
Inclusion Criteria:

* cvm stage 2-3
* mild to moderate class 2 mal occlusion
* no prior orthodontic treatment
* good oral hygiene
* good patient compliance

Exclusion Criteria:

* previous orthodontic treatment
* craniofacial anomlies
* severe crowding
* severe skeletal protrusion
* tmj disorders
* poor compliance
* dental anomales

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
improvement in ANB angle measured on lateral cephalometric radiographs (degrees) | 4-5 months

SECONDARY OUTCOMES:
changes in posterior airway space measured in mm using cbct | 4 -5 months
changes in TMJ measured in mm using cbct | 4-5 months

IPD SHARING:
Plan to Share IPD: Undecided